CLINICAL TRIAL: NCT00018213
Title: Naltrexone and Nicotine Replacement Effects on Cue Reactivity of Smokers
Brief Title: Naltrexone and Patch for Smokers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: ADRD-020-97F
Record Dates: First submitted 2001-07-03; First posted 2001-07-05 (Estimated); Last update posted 2009-01-21 (Estimated); Status verified 2007-09

CONDITIONS: Smoking
Keywords: Naltrexone; Nicotine patch; Tobacco dependence
MeSH Terms: conditions — Smoking; Tobacco Use Disorder | interventions — Naltrexone; Tobacco Use Cessation Devices

INTERVENTIONS:
Drug: Naltrexone Hydrochloride
Drug: Transdermal Nicotine

SUMMARY:
The aim of this study is to investigate the effects of naltrexone, alone and combined with nicotine patch, on responses of smokers to smoking cues after 10 hours of tobacco deprivation. Smokers who are not seeking treatment will be assigned to one of six conditions: They will receive either 50 mg of naltrexone or a placebo pill, and also will wear a nicotine patch that has 0, 21, or 42 mg of nicotine during the tobacco deprivation period. Both the day before the medication and deprivation and at the end of 10 hours of deprivation all will be exposed to lit cigarette cues in the laboratory. Effects of the medications will be assessed on withdrawal measures, urge to smoke, psychophysiological measures, and the topography of smoking three test cigarettes. Studies such as these can help to identify potential interventions for tobacco cessation or withdrawal, and thereby could result in less suffering and mortality.

ELIGIBILITY:
Adults who have smoked at least 25 cigarettes per day for at least a year. They are not using any method to quit smoking and are not using naltrexone. Must weigh at least 100lbs with no medical contraindications for naltrexone or transdermal nicotine. No contraindicated medications, no recent opiate use or history

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Dates: Start 1998-04; Study Completion 2001-03

CONTACTS AND LOCATIONS:
Locations (1):
- VA Medical Center, Providence, Rhode Island, United States